CLINICAL TRIAL: NCT00488800
Title: A Postmarketing Surveillance Study Evaluating the Safety and Local Tolerance of PREVENAR in Indian Children
Brief Title: Safety and Local Tolerability of Prevenar in Indian Children
Status: Completed | Type: Observational
Sponsor: Wyeth is now a wholly owned subsidiary of Pfizer (Industry)
Other Study IDs: 0887X-102324
Record Dates: First submitted 2007-06-18; First posted 2007-06-20 (Estimated); Last update posted 2007-12-28 (Estimated); Status verified 2007-12

CONDITIONS: Pneumococcal Infections
Keywords: Pneumococcal Infections/PC (Prevention & Control)
MeSH Terms: conditions — Pneumococcal Infections | interventions — Pneumococcal Vaccines

STUDY DESIGN:
Time Perspective: Prospective

INTERVENTIONS:
Biological: pneumococcal conjugate vaccine

SUMMARY:
This postmarketing surveillance study will evaluate the safety profile of Prevenar in Indian children.

Prevenar is indicated for active immunization of infants and children from 6 weeks of age through 9 years of age against invasive disease (including meningitis, bacteraemic pneumonia, bacteraemia, sepsis) caused by Streptococcus pneumoniae serotypes 4, 6B, 9V, 14, 18C, 19F and 23F.

Prevenar has been marketed in India since June 2006. The Board of Health in India has given restricted permission to import and market Prevenar. The present study is a post-approval regulatory commitment to the Board of Health in India.

This is an observational study and the protocol for the study has been approved by the Board of Health.

ELIGIBILITY:
INCLUSION CRITERIA

Subjects must meet at least one of the following conditions to be eligible for inclusion in the study:

For Primary Immunization Schedule:

* Healthy male or female subjects 6 weeks + 5 days of age with no previous PREVENAR vaccination
* For Catch-up Immunization Schedule:
* Healthy male or female subjects 12-23 months of age

EXCLUSION CRITERIA Subjects with any of the following conditions or characteristics will be excluded from the study.

* A known or suspected history of Streptococcus pneumoniae disease.
* A previous anaphylactic or other severe vaccine-associated adverse event.
* A known or suspected impairment of immune system (including HIV infection), or recipient of immunosuppressive agents.
* A major congenital, developmental or serious chronic disorder.
* A confirmed or suspected underlying evolving neurological disorder or history of seizures.
* A history of thrombocytopenia or any coagulation disorder.
* Any acute illness at the time of vaccine administration

Ages: 6 Weeks to 24 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 1000
Dates: Start 2006-07; Primary Completion 2007-01 (Actual); Study Completion 2007-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Wyeth is now a wholly owned subsidiary of Pfizer